CLINICAL TRIAL: NCT07107932
Title: A Large-Sample Real-World Dynamic Cohort Registry: Observing the Clinical Outcomes of Siltartoxatug Injection for Tetanus Prophylaxis Following Injury
Brief Title: A Registry： Siltartoxatug Injection for Tetanus Prophylaxis Following Injury
Status: Recruiting | Type: Observational
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TNM002-402
Record Dates: First submitted 2025-07-28; First posted 2025-08-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Tetanus
Keywords: Tetanus Prophylaxis
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Siltartoxatug Injection (Brand name: Sintetol®)
  Interventions: Drug: Siltartoxatug Injection (Brand name: Sintetol®)

INTERVENTIONS:
Drug: Siltartoxatug Injection (Brand name: Sintetol®) — The injury and wound conditions of the enrolled patients will be documented. A follow-up at 90 days post-administration will determine the clinical outcome of tetanus prophylaxis, specifically whether tetanus occurred. The registry will also employ selective safety data collection to record adverse reactions and serious adverse events following Siltartoxatug adminstration.

SUMMARY:
The injury and wound conditions of the enrolled patients will be documented. A follow-up at 90 days post-administration will determine the clinical outcome of tetanus prophylaxis, specifically whether tetanus occurred. The registry will also employ selective safety data collection to record adverse reactions and serious adverse events following Siltartoxatug adminstration.

ELIGIBILITY:
Inclusion Criteria:

* 1.Having received or will receive Siltartoxatug for tetanus prophylaxis following injury;
* 2. Provided signed informed consent by themselves or their legal representatives.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving Siltartoxatug for tetanus prophylaxis following injury and providing informed consent for participation.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | within 90 days
  Tetanus protection rate within 90 days post-administration of Siltartoxatug Injection (calculated as 1- tetanus incidence rate)

SECONDARY OUTCOMES:
Secondary Outcome | within 90 days
  Classification of wound characteristics in patients receiving Siltartoxatug Injection
Secondary Outcome | within 90 days
  Incidence of adverse reactions and serious adverse events within 90 days post-administration of Siltartoxatug Injection

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Second Affiliated Hospital of Shantou University, Shantou, Guangdong
  - Xiangyun County People's Hospital, Xiangyun, Yunnan
  - Shaoxing Central Hospital, Shaoxing, Zhejiang
  - Zhoushan Putuo District People's Hospital, Zhoushan, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided